CLINICAL TRIAL: NCT04018924
Title: Multi-center Study on the Effectiveness of Treatment With a Blue Light Medical Device (EmoLED) in Reduction of the Ulcer Surface in 10 Weeks
Brief Title: Blu Light for Ulcers Reduction
Acronym: BLUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emoled (Industry)
Collaborators: Akros Bioscience (Industry); Phidea Group (Industry); Istituto di Fisiologia Clinica CNR (Other); University of Pisa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EmoLED_002
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-03

CONDITIONS: Leg Ulcers Venous; Dehiscence, Surgical Wound
Keywords: Blue Light; Photo-bio-modulation; ulcers; leg ulcers Venous; dehiscence surgical wound; non healing wound
MeSH Terms: conditions — Varicose Ulcer; Surgical Wound Dehiscence; Ulcer | interventions — Ultraviolet Therapy

STUDY DESIGN:
Intervention Model Description: Patient used as control of himself: If a patient carries a wound with a diameter larger than 5 cm the wound is divided in two parts on treated with the Device the other covered and used as control, if the patient has two or more separate wounds each smaller than 5 cm in diameter the worst of them is treated the others used as control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T - Treated (Experimental): After standard cleansing or debridement of all wounds, on wound or portion of wound selected for treatment is treated with EmoLED device. Then covered with hydro fibre medication and dressing or compressive dressing when needed on the whole wound (SOC). Treatment is repeated once a week.
  Interventions: Device: Illumination with blue light (400-430nm) for 60 seconds with a power density of 120mW/sqcm (EmoLED device)

INTERVENTIONS:
Device: Illumination with blue light (400-430nm) for 60 seconds with a power density of 120mW/sqcm (EmoLED device) — Debridement and Dressing or compressive dressing if needed
  Other Names: Standard of Care (SOC)

SUMMARY:
Multi-center study on the effectiveness of treatment with a blue light medical device (EmoLED) in the reduction of ulcer surface in 10 weeks.

The aim of BLUR clinical trial is to verify if the proposed treatment represents a valid and significant remedy for Chronic Venous Insufficiency ulcers. The effectiveness will be measured through the evaluation of the reduction percentage of the lesion area during 10 weeks of treatment comparing the lesion (or portion of it) treated with EmoLED versus the control lesion (or portion of it) treated only according to current Standards of Care(SOC).

In the 10 weeks following the recruitment, the patient continues to follow the usual topical therapy with a frequency of once a week visit. The patient will be monitored up to the first event occurring: Complete healing or ten weeks. During the study, reports and evaluations will be made by medical staff on the device safety and usability.

90 patients will be recruited corresponding to the following criteria:

* Subjects suffering from venous, arterial and mixed skin ulcers and surgical dehiscence lesions;
* Presence of similar multiple lesions or lesions larger than 5 cm ;
* Men and women ≥ 18 years old;
* The patient must be able to understand the aims of the clinical study and provide informed consent in writing;
* Chronicity of the lesion: at least 8 weeks. The present clinical trial will be a multi-center prospective, controlled study with the aim of verifying the clinical efficacy of a portable battery-powered device based on blue LEDs.

We expect to record at least 20% of the difference between treated lesion and untreated lesion on the same patient during observation time.

The treatment, additional to the standard therapy for the patient, will be performed at each visit for 60 seconds on each 5 cm diameter sub-area of the selected lesion or on part of it.

In case of multiple lesions, one will be treated with EmoLED and one will be selected as a control lesion. In case of a very extensive lesion, it will be divided into two and one half will be the control of the other.

All lesions will be cleansed with saline solution and a surgical debridement will be performed with a scalpel if a slough/black base is present. Only then the treatment with EmoLED will begin.

If the patient has more than one lesion at the recruitment time, and all lesions are less than 5 cm in diameter, the worst lesions will be treated entirely with the EmoLED device and the others will constitute the control lesions. The evolution of all lesions in the ten weeks of the study duration will be evaluated.

If the patient has only one lesion greater than 5 cm in diameter at the recruitment time, the lesion will be divided into two parts along the major side and one half of the lesion area will be treated. The other half of the lesion will be masked with multi-layered sterile gauze during treatment. The point of division of the lesion into two parts will be indicated with an indelible marker and retouched at each visit.

If, at the time of recruitment, the patient has more than one lesion with a diameter greater than 5 cm, all lesions will be divided into two along the major side and will be treated as in the previous case.

After treatment with EmoLED, a hydrofiber dressing will be applied to the lesion. If clinical signs of infection occur, a hydrofiber dressing with silver will be applied. If necessary, compressive bandage of the limb will be carried out.

DETAILED DESCRIPTION:
A total of 90 subjects will be recruited at the facilities involved in the clinical study. All patients, both hospitalised and outpatient, will be considered for inclusion in this study.

The patients will be using a standard procedure that includes the evaluation of anamnesis and a physical examination.

All inclusion and exclusion criteria must be satisfied before recruitment. Any concomitant pharmacological therapy must be maintained.

Patients recruitment and screening The Principal Investigator or his delegate selects the enrolled patients on the basis of the inclusion and exclusion criteria of the study. Once the patient's correspondence with the study's criteria has been verified, the Principal Investigator or his delegate asks the patient for consent to use the EmoLED treatment device, and briefly explains the characteristics of the device and the expected effect. If the patient agrees, the Principal Investigator or his delegate proceeds to treatment. The patient must give his readiness to return to the structure every week for the established observation time.

Patient Identification Register The Principal Investigator is responsible for the updating and custody of the Patient Identification Register.

The Patient Identification Register contains the personal data of the patients participating in the study, the date of recruitment and the patient code (the structure number followed by a progressive two-digit numerical code).

Only the Principal Investigator and, at the discretion of the Principal Investigator, the members of his team know the identity of the patients enrolled in the study.

If a patient withdraws from the study, the Principal Investigator or his delegate records the event in the Patient Identification Register and on the Data Collection Form and stores all documentation.

Patient Enrolment Format For each new patient, the Principal Investigator or his delegate fills the Patient Enrolment Format that contains data such as patient identification (Name and Surname are to be understood as those of the data collection form, ie identification code of the center and number), age, gender, aetiology of the ulcer, any concomitant diseases, drug therapy, date of ulcers beginning and date of recruitment.

The second part of the format contains a table in which the date of the visit, the data on the patient's health, and the data collected are recorded at each visit.

Registration of clinical data The data related to the evaluation of the study endpoints are acquired at precise times, corresponding to the timepoints reported in the protocol and in the Data Collection Form.

The parameters of the Data Collection Form are acquired and maintained on paper format for the duration of the trial. Once the study on the patient has been completed, they are kept in both paper and digital format, after scanning the paper form. The photos of the wound are acquired and stored in digital format, both for the duration of the study and subsequently.

Data Collection Form The Data Collection Form is unique for each patient. It consists of some columns to fill in according to the observation times. At each visit, the doctor indicates with an "X" the value chosen for each parameter.

The Data Collection Form is scanned and archived after the patient's discharge or withdrawal of the trial.

Centralised database The Principal Investigator sends to the Project Manager the Patient Enrolment Formats of the new recruited patients and the photographic records of the all patients returned to the control every week. For patients leaving the study, the Data Collection Form will also be transmitted.

The Project Manager creates a unique database of all the patients, updated every week with the latest available data and consulted by the Principal Investigators. The creation of this database allows investigators to be aware of the number of patients still to be recruited and of the study progress.

Data recording Following the recruitment and the signing of the informed consent, the data relevant to each patient will be collected in the Data Collection Form at different times: S0 (Week 0: recruitment and first treatment), S1, S2, S3 ... up to S10 (visits in the 10 weeks following recruitment).

Patients may miss a maximum of two not consecutive visits, starting from the fifth visit. The patient who misses one of the first four visits or two consecutive visits, will be excluded from the study.

The parameters used to define the study result will be found through:

* photographic images of lesions treated with EmoLED and control lesions
* Data Collection Form filled by the personnel during the visit.

SERIOUS ADVERSE EVENTS (SAE) Although the available literature and the in vivo tests performed provide reasonable certainty of the safety of the device in case of the occurrence of SAE it will be managed according to the following procedures: Good Clinical Practice Med Dev 2.7/3 and International Standard Organisation 14155. There will be a constant monitoring of the health condition of the patient during the trial phase and for a reasonable period of time after the trial end. Any SAE reported by the patient and/or the investigator or any member of his team will be reported through the module "Adverse Event Module" and timely communicated to the Competent Authority.

CALCULATION OF SAMPLE NUMEROSITY The choice of the statistical model used is based on the literature research on wound healing trends and the past clinical experience and recorded data of the hospital center involved in the study. The most relevant information emerged is that at 10 weeks is expected a 30% variability in the reduction percentage of the wound dimension. This value is confirmed by [15 see citation] where has been used for the sample sizing. Moreover in [16 see citation] a 53% deviation standard of the lesion reduction percentage in the worst case of venous ulcers.

The analysis for the sample sizing is based upon:

The clinical goal expressed in the percentage of reduction of the lesion area at ten weeks; The non-parametric statistical test for pair of data, consisting in the Wilcoxon rank-sum test; An a priori hypothesis of 50% on the expected variability (conservative value); An average 20% difference between treated and non-treated; A statistical power equal to 80% (Beta=0.2) and Afa =0.05; The unilateral alternative hypothesis: the EmoLED treatment does not worsen the outcome; A correlation coefficient between treated area versus non treated area equal to 0.1, 0.3, 0,5 and 0.7; The numerosity of the sample is calculated according to the method of the relative asymptotic efficiency in respect to the t test (min AREA), the case of R =0.1 (minimum coefficient) indicate N=83 patients , this has been used to establish in 90 patients the sample numerosity (considering the drop out risk).

Statistical analysis of the primary endpoint The device effectiveness will be measured performing a Wilcoxon signed rank test with a one-sided level of significance Alfa=0.05. This test is useful for analysing paired data and takes in to consideration the sign and the magnitude of the observed differences. There will be an analysis of the entire protocol as well as of different possible populations.

STATISTICAL ANALYSIS OF THE SECONDARY ENDPOINT

1. Safety: all SAE recorded will be managed with the appropriate statistical instrument according to the size and type of events reported.
2. Comparison of the outcome in terms of percentage reduction of the wound treated with EmoLED + SOC versus the one treated only with SOC in the 10 weeks of observation: At every observation date both treated and non-treated wound will be measured. The pair data will be statistically analysed with repeated measures. There will be both a punctual analysis as well as an overall trend analysis of the whole period considered. In the first case the paired data will be observed using a parametric test (t-test) or a non-parametric test (Wilcoxon of the signed rank) according to the data distribution observed. A correction of the statistical significance such as the Benjamini-Hochberg correction will be applied. In the second case, a view of the differences in healing trends between treated and non- treated will be obtained through the evaluation of the are under the curve for each subject an in each area. The paired data will be observed using a parametric or a non-parametric test. In both cases, missing data will be replaced using the mean value of the other patients. A sensitivity analysis will be performed using the max and min value observed in patients.
3. Evaluation of the gap in healing time between the two areas: A survival analysis based on the Akritas test applied to the Kaplan-Meier curves will be used. Such analysis is useful to evaluate the time to reach the event of interest that in this case is reaching healing level > or = to 70% in 10 weeks. Such technique can handle paired data and the event of possible drop outs. For each group (treated and non-treated) will be built a curve , the Akritas test is based on a transformation in ranks of the "survival" times intended as the "time to event" considered as a healing level > or = to 70% in 10 weeks. The ranks will be transformed according to a model that allows stop and censures.
4. Pain reduction measured with a Visual Analogical Scale (VAS) 0-10. A non-parametric Friedman test will be used, the equivalent of a non-parametric test ANOVA for repeated measures.

All data regarding the patients will be maintained as strictly confidential and their informed consensus obtained at the enrolment time will be identified with a coding system all investigator will keep the data up to two years after the study's end.

MONITORING The study coordination is assigned to an independent third party qualified for the purpose (independent CRO), it will be responsible for the adherence to the International Conference on Harmonization (ICH)/Good Clinical Practice (GCP) guidelines. The coordinator will perform regular monitoring visits at the investigator site to make sure that all data are properly recorded and maintained it will have access to all data to ensure the adherence to the Protocol and the accuracy, coherence and precision of the data collected.

ETHICAL CONSIDERATIONS The study will be submitted to the Ethical Committee of each investigator hospital for approval and in any case will be performed according to the Helsinki Declaration and the Italian laws and requirements in the matter of human clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from venous, arterial and mixed skin ulcers and surgical dehiscence lesions;
* Presence of similar multiple lesions or lesions larger than 5 cm ;
* The patient must be able to understand the aims of the clinical study and provide informed consent in writing;
* Chronicity of the lesion: at least 8 weeks.

Exclusion Criteria:

* Patients who participated in a clinical study on skin ulcers healing during the previous month;
* Patients who are unable to understand the aims and the objectives of the study;
* Patients with neoplastic ulcers;
* Patients with decubitus ulcers;
* Patients with diabet foot ulcers;
* Patients with infected ulcers;
* Patients with ulcers caused by critical ischemia;
* Patients with a past of self-harm that can purposely alter the progress of healing;
* Patients with psychiatric disorders;
* Pregnancy or breast feeding ;
* Patients with neoplasms or other diseases involving the use of cytostatic or immunosuppressive drugs;
* Patients with limited lifespan.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2019-11-17 (Actual); Study Completion 2019-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Fraccalvieri, Doctor, Principal Investigator — A.O.U. Città della Salute e della Scienza; Stefano Gasperini, Doctor, Study Director — Medical Advisor
Locations (7):
- Italy (7):
  - Ospedale Umberto I-Wound and Diabetic foot ambulatory, Bari
  - Barbantini Clinic, Lucca
  - Lucca Hospital, Lucca
  - Policlinico G. Martino, Messina
  - ASL Napoli 3 Sud, Naples
  - Saint Luca Clinic, Turin
  - San Lazzaro Hospital - Plastic Surgery Department, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mast BA, Schultz GS. Interactions of cytokines, growth factors, and proteases in acute and chronic wounds. Wound Repair Regen. 1996 Oct;4(4):411-20. doi: 10.1046/j.1524-475X.1996.40404.x. PMID 17309691
- [Background] Nwomeh BC, Yager DR, Cohen IK. Physiology of the chronic wound. Clin Plast Surg. 1998 Jul;25(3):341-56. PMID 9696897
- [Background] Hackam DJ, Ford HR. Cellular, biochemical, and clinical aspects of wound healing. Surg Infect (Larchmt). 2002;3 Suppl 1:S23-35. doi: 10.1089/sur.2002.3.s1-23. PMID 12573037
- [Background] Beani JC, Jeanmougin M. [Narrow-band UVB therapy in psoriasis vulgaris: good practice guideline and recommendations of the French Society of Photodermatology]. Ann Dermatol Venereol. 2010 Jan;137(1):21-31. doi: 10.1016/j.annder.2009.12.004. Epub 2009 Dec 29. French. PMID 20110064
- [Background] Adamskaya N, Dungel P, Mittermayr R, Hartinger J, Feichtinger G, Wassermann K, Redl H, van Griensven M. Light therapy by blue LED improves wound healing in an excision model in rats. Injury. 2011 Sep;42(9):917-21. doi: 10.1016/j.injury.2010.03.023. PMID 22081819
- [Background] Clark RA. Cutaneous tissue repair: basic biologic considerations. I. J Am Acad Dermatol. 1985 Nov;13(5 Pt 1):701-25. doi: 10.1016/s0190-9622(85)70213-7. PMID 2416789
- [Background] Son GY, Hong JH, Chang I, Shin DM. Induction of IL-6 and IL-8 by activation of thermosensitive TRP channels in human PDL cells. Arch Oral Biol. 2015 Apr;60(4):526-32. doi: 10.1016/j.archoralbio.2014.12.014. Epub 2014 Dec 25. PMID 25575297
- [Background] Bertin S, Aoki-Nonaka Y, de Jong PR, Nohara LL, Xu H, Stanwood SR, Srikanth S, Lee J, To K, Abramson L, Yu T, Han T, Touma R, Li X, Gonzalez-Navajas JM, Herdman S, Corr M, Fu G, Dong H, Gwack Y, Franco A, Jefferies WA, Raz E. The ion channel TRPV1 regulates the activation and proinflammatory properties of CD4(+) T cells. Nat Immunol. 2014 Nov;15(11):1055-1063. doi: 10.1038/ni.3009. Epub 2014 Oct 5. PMID 25282159
- [Background] Xu T, Wu BM, Yao HW, Meng XM, Huang C, Ni MM, Li J. Novel insights into TRPM7 function in fibrotic diseases: a potential therapeutic target. J Cell Physiol. 2015 Jun;230(6):1163-9. doi: 10.1002/jcp.24801. PMID 25204892
- [Background] Kleinpenning MM, Smits T, Frunt MH, van Erp PE, van de Kerkhof PC, Gerritsen RM. Clinical and histological effects of blue light on normal skin. Photodermatol Photoimmunol Photomed. 2010 Feb;26(1):16-21. doi: 10.1111/j.1600-0781.2009.00474.x. PMID 20070834
- [Background] Cicchi R, Rossi F, Alfieri D, Bacci S, Tatini F, De Siena G, Paroli G, Pini R, Pavone FS. Observation of an improved healing process in superficial skin wounds after irradiation with a blue-LED haemostatic device. J Biophotonics. 2016 Jun;9(6):645-55. doi: 10.1002/jbio.201500191. Epub 2016 Jan 12. PMID 26756549
- [Background] Rossi et al. (2010), A blue-LED-based device for selective photocoagulation of superficial abrasions: theoretical modeling and in vivo validation, Photonic Therapeutics and Diagnostics VI, Proceedings of SPIE Volume: 7548.
- [Background] Meaume S, Dissemond J, Addala A, Vanscheidt W, Stucker M, Goerge T, Perceau G, Chahim M, Wicks G, Perez J, Tacca O, Bohbot S. Evaluation of two fibrous wound dressings for the management of leg ulcers: results of a European randomised controlled trial (EARTH RCT). J Wound Care. 2014 Mar;23(3):105-6,108-11, 114-6. doi: 10.12968/jowc.2014.23.3.105. PMID 24633056
- [Background] Hansson C. The effects of cadexomer iodine paste in the treatment of venous leg ulcers compared with hydrocolloid dressing and paraffin gauze dressing. Cadexomer Iodine Study Group. Int J Dermatol. 1998 May;37(5):390-6. doi: 10.1046/j.1365-4362.1998.00415.x. PMID 9620490
- [Background] Marston WA, Carlin RE, Passman MA, Farber MA, Keagy BA. Healing rates and cost efficacy of outpatient compression treatment for leg ulcers associated with venous insufficiency. J Vasc Surg. 1999 Sep;30(3):491-8. doi: 10.1016/s0741-5214(99)70076-5. PMID 10477642
- [Background] F. Petrella, Progetto SIUC (Studio Incidenza Ulcere Cutanee), 1 gennaio 2015 - 31 dicembre 2016, AIUC
- [Background] M. Fraccalvieri "Le terapie della deiscenza dell'incisione chirurgica" Ediz Minerva Medica, pag 17, Aprile 2015, Torino, Italy, ISBN 9-788877-118325

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The total number of participants is 90 and the patient is control of himself.
Groups:
- All Participants: The patient is control of themselves so all participants received both interventions; for each patient are treated and evaluated two different wounds (or two different parts of wound).
  Control wound:
  After standard cleansing or debridement of all wounds, the wound is covered with hydro fibre medication and dressing or compressive dressing when needed on the whole wound (SOC). The medication and dressing are repeated once a week.
  EmoLED treated wound:
  After standard cleansing or debridement of all wounds, on wound or portion of wound selected for treatment is treated with EmoLED device. Then covered with hydro fibre medication and dressing or compressive dressing when needed on the whole wound (SOC). Treatment is repeated once a week.
  Illumination with blue light (400-430nm) for 60 seconds with a power density of 120mW/sqcm (EmoLED device).
Period: Overall Study
Arm/Group | All Participants
Started | 90 (The total number of participants is 90 and the patient is control of themselves.)
Standard Of Care Intervention | 90
EmoLED Intervention | 90
Completed | 84
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 90
Age, Customized [Count of Participants; unit: Participants]
  Age groups: < 49 years | 7
  Age groups: 50 < years < 59 | 12
  Age groups: 60 < years < 69 | 16
  Age groups: 70 < years < 79 | 28
  Age groups: 80 < years <89 | 26
  Age groups: > 90 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 90

OUTCOME MEASURES:

1. Primary Outcome: Size of Wound Remaining Compared to Initial Wound Size
Description: The primary outcome of the study is the outcomes comparison as remaining wound area surface percentage difference of the lesion treated with EmoLED versus the lesion treated with SOC, both as difference on same patient and within the group of all recruited patients.
  The primary outcome is measured as the average of the ratio between final areas and initial areas; the ratio of 10 week wound surface area to initial wound surface area was multiplied by 100 to determine the percentage.
Time Frame: 10 weeks
Population: Non-compliant and dropout patients were excluded. Only patients whose images could be analyzed were considered in the analysis.
Measure: Mean (Standard Deviation); unit: percentage of the remaining area
Arm/Group | All Participants
Number analyzed (Participants) | 67
percentage of the remaining area
  EmoLED treated wound | 42.58 (39.7)
  Control wound | 53.78 (84.8)

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: Presence of any Adverse event during treatment period and after
Time Frame: 10 weeks treatment or in case of adverse event until the patient status return to normal
Population: All Treatment-Emergent Adverse Events were systemic and cannot be attributed to one or the other intervention, due to the fact that all patients are also control of themselves.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 90
Participants | 6

3. Secondary Outcome: Weekly Comparison of Healing Percentage
Description: Outcomes comparison as percentage reduction of the lesion treated with EmoLED versus the lesion treated with SOC within ten weeks of the study. The measure of the outcome was calculated by the average of the medians of the weekly percentage reduction of the area, compared to the previous visit.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of area reduction
Arm/Group | All Participants
Number analyzed (Participants) | 67
percentage of area reduction
  EmoLED treated wound | 7.02 (4.19)
  Control wound | 3.06 (3.72)

4. Secondary Outcome: Percentage of Recovered Wounds at 10 Weeks
Description: Time difference measured in weeks to reach the healing. The analysis was conducted deriving the Kaplan-Meyer curves from the analysis of the healing time. The K-M curves describe the probability of healing at each control time.
Time Frame: 10 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of probability of recovery
Arm/Group | All Participants
Number analyzed (Participants) | 67
percentage of probability of recovery
  EmoLED treated wound | 24
  Control wound | 18

5. Secondary Outcome: Pain Change
Description: pre-treatment evaluation with Visual Analogic Scale (0-10 scale with 0 as no pain and 10 as extreme pain) and comparison with the same scale measured at each treatment. The result is measured by writing the averages of Week 1 and of Week 10.
Time Frame: Week 1 and Week 10
Population: The analysis was carried out considering the subjects who have 11 assessments, until yhe 10th week. The pain cannot be attributable to one or the other intervention because the patient is control of themselves, so pain cannot be perceived separately by the individual.
Measure: Number; unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 45
units on a scale
  Visit 0 | 7.2
  Visit 10 | 4.6

6. Secondary Outcome: Event of Recidivism
Description: At the discretion of the patient's willingness to continue to visit the study site; observation of the unhealed area(s) over the 10-week period is extended until healing or up to 20 weeks.
Time Frame: 20 weeks
Population: It was at the discretion of the patient's willingness to continue the observation time after the 10 weeks of treatment. None of the patients that presented an unhealed area over the 10-week period decided to continue.
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 15 months
Description: Adverse Events reported in this study cannot be attributed to one or the other intervention, due to the fact that they are systemic and all patients are also control of themselves.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 5/90
Other Adverse Events (participants affected / at risk) | 1/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=90)
POA with critical stenosis (Blood and lymphatic system disorders) | 1
Myocardial infarction and heart failure (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Hyperthermia/ Erysipelas (Skin and subcutaneous tissue disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=90)
Fistulae (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04018924/Prot_SAP_000.pdf